CLINICAL TRIAL: NCT06459739
Title: Effect of Sacral Erector Spinae Plane Block on Hemorrhoid and Pilonidal Sinus Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Erzincan Binali Yildirim Universitesi (Other)
Responsible Party: Principal Investigator, Alparslan Koc, Assoc. Prof., Erzincan Binali Yildirim Universitesi
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: SacralESPB
Record Dates: First submitted 2024-06-05; First posted 2024-06-14 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Pain, Acute Post-Operative; Pilonidal Sinus; Hemorrhoids; Anesthesia
Keywords: Sacral ESPB; Postoperative pain; Hemorrhoidectomy; Pilonidal sinus surgery; Analgesia
MeSH Terms: conditions — Pain, Postoperative; Pilonidal Sinus; Hemorrhoids; Agnosia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- sacralESPB (Experimental): Sacral ESPB group
  Interventions: Procedure: sacral ESPB
- Control (No Intervention)

INTERVENTIONS:
Procedure: sacral ESPB — sacral ESPB
  Arms: sacralESPB

SUMMARY:
Introduction: This study investigated the efficacy of sacral erector spinae plane block (ESPB) for managing postoperative pain and reducing opioid consumption in patients undergoing hemorrhoid and pilonidal sinus (PS) surgery.

DETAILED DESCRIPTION:
Introduction: This study investigated the efficacy of sacral erector spinae plane block (ESPB) for managing postoperative pain and reducing opioid consumption in patients undergoing hemorrhoid and pilonidal sinus (PS) surgery.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) I-II patients undergoing hemorrhoid and pilonidal sinus surgery

Exclusion Criteria:

* patients with coagulopathies, pregnant women, patients with significant cardiovascular, hepatic, or renal disease, patients who declined spinal anesthesia or were contraindicated for it, and patients who had previously undergone the same surgery

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-04-01 (Actual)

PRIMARY OUTCOMES:
Postoperative pain | 0.5,2,8,24 hours
  Numeric rating scale evaluation after surgery. Use 0 to 10 points with 0 no pain 5 moderate pain and 10 severe pain.

SECONDARY OUTCOMES:
Opioid consumption | 0.5,2,8,24 hours
  Admission of tramadol as a rescue analgesia

CONTACTS AND LOCATIONS:
Locations (1):
- Erzincan Binali Yildirim university, Erzincan, Turkey (Türkiye)